CLINICAL TRIAL: NCT01069536
Title: Efficacy and Akathisia Incidence of Slow Infusion Metoclopramide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PAU-200/030-0515
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2007-03

CONDITIONS: Akathisia; Nausea
Keywords: metoclopramide; akathisia; nausea; vomiting; antiemetic; improvement of nausea
MeSH Terms: conditions — Psychomotor Agitation; Nausea; Vomiting | interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 2 minutes bolus infusion (Active Comparator)
  Interventions: Drug: metoclopramide 10 mg
- 15 minutes slow infusion (Active Comparator)
  Interventions: Drug: metoclopramide 10 mg

INTERVENTIONS:
Drug: metoclopramide 10 mg

SUMMARY:
Study Objective:

The purpose of this study is to compare the effects of metoclopramide administration in bolus versus slow infusion medications in ED patients complaining of nausea for the determination of the therapeutic effect and prevention of akathisia.

Methods:

This was a prospective, randomized, double-blind trial. The investigation was held between 01 March 2007 and 01 May 2008, in the Emergency Department of Pamukkale University Faculty of Medicine. The patients with moderate to severe nausea randomized and divided into two groups as for the previously planned administration type of drug. Ten mg metoclopramide was administered in one group with slow infusion (SIG) in 15 minutes, via 2 minutes bolus infusion (BIG) into the other group. Whole procedure was observed, akathisia and nausea scores and vital changes were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 through 65 years of age and 50-90 kg of weight who presented to the ED with primary or secondary complaints of moderate to severe nausea who not use of commonly accepted antiemetic within the previous 24 hours were eligible for this study.
* Their peripheral oxygen saturation level was 90% or over while respirating room air and free of any respiratory problems.

Exclusion Criteria:

* Patients with mild symptoms of nausea
* Altered mental status
* Abnormal vital signs
* Any known allergy to the metoclopramide
* Previously enrolled in the study
* Known renal failure or insufficiency
* GIS hemorrhage, ileus and/or perforation
* Women who were pregnant and lactating
* Those with a history of epilepsy
* Admitted to the ED due to acute psychiatric symptoms
* Restless legs syndrome
* Parkinson
* Organic brain disease
* Phaeochromocytoma
* Patient with alcohol
* Anticholinergic, sedative, hypnotic, trankilizan, digoxin, cimetidine, tetracycline and levo-dopa use
* Presence of severe agitation akathisia can not be evaluated and uncooperative individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-03; Primary Completion 2007-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
akathisia and nausea scores